CLINICAL TRIAL: NCT01577810
Title: Near Infrared Spectroscopy (NIRS) for Heart Failure Assessment in the Outpatient Setting
Brief Title: Near Infrared Spectroscopy (NIRS) for Heart Failure Assessment.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigator did not have appropriate time to complete the study.
Sponsor: Phoenix Children's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PHNX-NIRS-12-024
Record Dates: First submitted 2012-03-23; First posted 2012-04-16 (Estimated); Last update posted 2025-11-24 (Actual); Status verified 2017-04

CONDITIONS: Cardiac Failure
Keywords: NIRS; near infrared spectroscopy; heart failure; cardiac output; outpatient; pediatric
MeSH Terms: conditions — Heart Failure | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Intervention Model Description: The NIRS monitoring in the heart center was not able to be completed.
Masking Description: Only the investigator knew the assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- non-NIRS patients (Other)
  Interventions: Device: Near Infrared Spectroscopy

INTERVENTIONS:
Device: Near Infrared Spectroscopy — Use of Near Infrared Spectroscopy in outpatient setting to determine global cardiac output
  Other Names: NIRs; INVOS

SUMMARY:
It is routine practice for a cardiologist to perform a battery of tests to assess the degree of heart failure. The purpose of this study is to establish a non-invasive method to reliably predict cardiac output state in real-time in children and adolescents with heart failure in an outpatient setting. This study will rely on the use of near infrared spectroscopy monitors to measure cardiac output in the outpatient setting.

DETAILED DESCRIPTION:
Near-infrared spectroscopy (NIRS) technology, such as that used in pulse oximetry, has been used in medicine for decades. Several characteristics contribute to its widespread use, including its noninvasive nature, reliability and safety. The Somanetics' INVOS® System harnesses this power to safely and reliably "see inside" the brain and body. NIRS devices measure the venous weighted oxy-hemoglobin saturation (color of blue blood) in a field of tissue, rather than in arteries, and thus the rSO2 parameter provides a window into regional oxygen supply-demand relationships. Monitoring rSO2 at two distinct sites (cerebral and somatic) has become common practice at our institution for all infants and children in the intensive care unit and provides valuable feedback about potentially deleterious trends in regional tissue oxygenation that cannot easily be obtained by other modalities in such patients.

ELIGIBILITY:
Inclusion Criteria:

* Patient in Phoenix Children's Hospital Heart Failure Clinic

Exclusion Criteria:

* N/A

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2013-06; Primary Completion 2017-04-05 (Actual); Study Completion 2017-04-05 (Actual)

PRIMARY OUTCOMES:
Degree of Heart Failure using NIRS | 5 minutes
  The investigators strive to discover a surrogate marker for uncompensated heart failure. The use of two-site NIRS monitoring for global cardiac output assessment, through the patterning of somatic and cerebral saturation data in combination with pulse-oximetry data and other vital signs in the outpatient setting, has not been researched although it is used widely in the inpatient arena.

CONTACTS AND LOCATIONS:
Overall Officials: Rohit Rao, MD, Principal Investigator — Phoenix Children's Hospital
Locations (1):
- Phoenix Children's Hospital Heart Failure Clinic, Phoenix, Arizona, United States

REFERENCES:
- [Background] Hayashida M, Kin N, Tomioka T, Orii R, Sekiyama H, Usui H, Chinzei M, Hanaoka K. Cerebral ischaemia during cardiac surgery in children detected by combined monitoring of BIS and near-infrared spectroscopy. Br J Anaesth. 2004 May;92(5):662-9. doi: 10.1093/bja/aeh120. Epub 2004 Mar 19. PMID 15033888
- [Background] Hoffman GM, Stuth EA, Jaquiss RD, Vanderwal PL, Staudt SR, Troshynski TJ, Ghanayem NS, Tweddell JS. Changes in cerebral and somatic oxygenation during stage 1 palliation of hypoplastic left heart syndrome using continuous regional cerebral perfusion. J Thorac Cardiovasc Surg. 2004 Jan;127(1):223-33. doi: 10.1016/j.jtcvs.2003.08.021. PMID 14752434
- [Background] Nollert G, Jonas RA, Reichart B. Optimizing cerebral oxygenation during cardiac surgery: a review of experimental and clinical investigations with near infrared spectrophotometry. Thorac Cardiovasc Surg. 2000 Aug;48(4):247-53. doi: 10.1055/s-2000-6895. PMID 11005605
- [Background] Watzman HM, Kurth CD, Montenegro LM, Rome J, Steven JM, Nicolson SC. Arterial and venous contributions to near-infrared cerebral oximetry. Anesthesiology. 2000 Oct;93(4):947-53. doi: 10.1097/00000542-200010000-00012. PMID 11020744
- [Background] Wyatt JS, Cope M, Delpy DT, Wray S, Reynolds EO. Quantification of cerebral oxygenation and haemodynamics in sick newborn infants by near infrared spectrophotometry. Lancet. 1986 Nov 8;2(8515):1063-6. doi: 10.1016/s0140-6736(86)90467-8. PMID 2877225
- [Background] Yoshitani K, Kawaguchi M, Iwata M, Sasaoka N, Inoue S, Kurumatani N, Furuya H. Comparison of changes in jugular venous bulb oxygen saturation and cerebral oxygen saturation during variations of haemoglobin concentration under propofol and sevoflurane anaesthesia. Br J Anaesth. 2005 Mar;94(3):341-6. doi: 10.1093/bja/aei046. Epub 2004 Dec 10. PMID 15591331
- [Background] Fortune PM, Wagstaff M, Petros AJ. Cerebro-splanchnic oxygenation ratio (CSOR) using near infrared spectroscopy may be able to predict splanchnic ischaemia in neonates. Intensive Care Med. 2001 Aug;27(8):1401-7. doi: 10.1007/s001340100994. PMID 11511955
- [Background] Petros AJ, Heys R, Tasker RC, Fortune PM, Roberts I, Kiely E. Near infrared spectroscopy can detect changes in splanchnic oxygen delivery in neonates during apnoeic episodes. Eur J Pediatr. 1999 Feb;158(2):173-4. doi: 10.1007/s004310051046. No abstract available. PMID 10048622
- [Background] Nagdyman N, Fleck T, Barth S, Abdul-Khaliq H, Stiller B, Ewert P, Huebler M, Kuppe H, Lange PE. Relation of cerebral tissue oxygenation index to central venous oxygen saturation in children. Intensive Care Med. 2004 Mar;30(3):468-71. doi: 10.1007/s00134-003-2101-8. Epub 2004 Jan 13. PMID 14722637
- [Background] Schulz G, Weiss M, Bauersfeld U, Teller J, Haensse D, Bucher HU, Baenziger O. Liver tissue oxygenation as measured by near-infrared spectroscopy in the critically ill child in correlation with central venous oxygen saturation. Intensive Care Med. 2002 Feb;28(2):184-9. doi: 10.1007/s00134-001-1182-5. Epub 2002 Jan 12. PMID 11907662
- [Background] Weiss M, Dullenkopf A, Kolarova A, Schulz G, Frey B, Baenziger O. Near-infrared spectroscopic cerebral oxygenation reading in neonates and infants is associated with central venous oxygen saturation. Paediatr Anaesth. 2005 Feb;15(2):102-9. doi: 10.1111/j.1460-9592.2005.01404.x. PMID 15675925
- [Background] Nollert G, Mohnle P, Tassani-Prell P, Uttner I, Borasio GD, Schmoeckel M, Reichart B. Postoperative neuropsychological dysfunction and cerebral oxygenation during cardiac surgery. Thorac Cardiovasc Surg. 1995 Oct;43(5):260-4. doi: 10.1055/s-2007-1013224. PMID 8610284
- [Background] Berens RJ, Stuth EA, Robertson FA, Jaquiss RD, Hoffman GM, Troshynski TJ, Staudt SR, Cava JR, Tweddell JS, Bert Litwin S. Near infrared spectroscopy monitoring during pediatric aortic coarctation repair. Paediatr Anaesth. 2006 Jul;16(7):777-81. doi: 10.1111/j.1460-9592.2006.01956.x. PMID 16879521
- [Background] Tsuji M, Saul JP, du Plessis A, Eichenwald E, Sobh J, Crocker R, Volpe JJ. Cerebral intravascular oxygenation correlates with mean arterial pressure in critically ill premature infants. Pediatrics. 2000 Oct;106(4):625-32. doi: 10.1542/peds.106.4.625. PMID 11015501
- [Background] Hanson SJ, Berens RJ, Havens PL, Kim MK, Hoffman GM. Effect of volume resuscitation on regional perfusion in dehydrated pediatric patients as measured by two-site near-infrared spectroscopy. Pediatr Emerg Care. 2009 Mar;25(3):150-3. doi: 10.1097/PEC.0b013e31819a7f60. PMID 19262423
- [Background] Bernal NP, Hoffman GM, Ghanayem NS, Arca MJ. Cerebral and somatic near-infrared spectroscopy in normal newborns. J Pediatr Surg. 2010 Jun;45(6):1306-10. doi: 10.1016/j.jpedsurg.2010.02.110. PMID 20620336